CLINICAL TRIAL: NCT05282966
Title: Assessment of QSant™ for Underlying Allograft Rejection (AQUA Registry)
Brief Title: Assessment of QSant™ for Underlying Allograft Rejection
Acronym: AQUA
Status: Not yet recruiting | Type: Observational
Sponsor: NephroSant (Industry)
Responsible Party: Sponsor
Other Study IDs: NEPHRO-001
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: kidney transplant; kidney biopsy; allograft rejection; subclinical allograft rejection; kidney; kidney health; kidney function; urine sample; urine test; kidney disease
MeSH Terms: conditions — Rejection, Psychology; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Cohort with QSant Testing: 2,000 participants will be enrolled across sites within 90-days post-kidney transplant and followed for 24-months
  Interventions: Diagnostic Test: QSant-TM Urine Test
- Retrospective Control Cohort without QSant Testing: 2,000 site-matched controls from UNOS database who underwent a kidney transplant no more than 5 years prior to the study completion date

INTERVENTIONS:
Diagnostic Test: QSant-TM Urine Test — QSant™ is a needle free urine test collected in-home or in-clinic to aid in the evaluation and management of kidney transplant recipients' allograft status. QSant evaluates 6 kidney-specific biomarkers.
  Other Names: QSant(TM); QScore(TM)
  Groups: Prospective Cohort with QSant Testing

SUMMARY:
The AQUA registry is a multi-center observational study to assess the clinical management of kidney transplant recipients (KTRs) with use of the QSant test. QSant is a test based on 6 urinary biomarkers including cell-free DNA, that is used for the evaluation and management of acute rejection in renal allograft recipients with clinical suspicion of rejection, as well as subclinical rejection.

DETAILED DESCRIPTION:
The AQUA registry is a multi-center observational study to assess the clinical management of kidney transplant recipients (KTRs) with use of the QSant test. Each participant will be tracked for 24 months. QSant testing will be performed according to the intended use guidelines specified in "LCD - MolDX: Molecular Testing for Solid Organ Allograft Rejection (L38671)", along with all standard of care testing, such as serum creatinine/ estimated glomerular filtration rate (SCr/eGFR) as described in the study schedule. Participants will be compared to a site-specific retrospective cohort of KTRs without QSant testing having received a kidney transplant no more than 5 years prior to study initiation as well as the national cohort derived from UNOS (United Network for Organ Sharing) data.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant recipient, ≤ 90 days post kidney transplant of any age, solitary or combined multi-organ solid transplants which includes a kidney transplant.
2. Able to understand risks and requirements of participation and provide informed consent
3. Willing and able to comply with the study requirements

Exclusion Criteria:

1. Inability to provide a voided urine sample per collection protocol
2. Urological abnormalities such as augmented bladder, ileo-conduits, mitrofanoff, and vesicostomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients of all ages
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
QScore specificity and sensitivity in relation to kidney biopsy | 6 weeks before each biopsy-proven rejection (BPAR)
  Demonstrate sensitivity and specificity of QSant for detecting biopsy-proven rejection (BPAR), defined as t-score ≥1. For this aim QSant detection will be based on a threshold of >32 within 6 weeks of BPAR (using the most recently collected result)